CLINICAL TRIAL: NCT02901249
Title: Assessment of Cost- Effectiveness Interventions and the Quality of Life in Patients With Major Depression Through Resources Available in Brazilian Public Health
Brief Title: Cost- Effectiveness and Quality of Life Assessment in Major Depression Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federal University of Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Ana Flávia Barros da Silva Lima, Principal Investigator, Federal University of Rio Grande do Sul
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 017/2009
Record Dates: First submitted 2016-09-11; First posted 2016-09-15 (Estimated); Results first posted 2020-10-14 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2016-08

CONDITIONS: Depression
Keywords: Cost effectiveness; Unipolar Depression; Major Depression Disorder; Quality of life disorder
MeSH Terms: conditions — Depression; Depressive Disorder | interventions — Sertraline; Nortriptyline; Lithium; Lithium Carbonate

STUDY DESIGN:
Intervention Model Description: Patients start treatment according to the algorithm and follow a sequence of steps. There is no comparison between groups. It is a single group. Primary and secondary outcomes are only assessed at the end of the protocol, not at each step.
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sertraline (Experimental): Group Started: sertraline (50mg-200mg)
  Subjects evaluated for responsiveness every 2 weeks. Responsive to treatment patients remain in the same step. Max. step duration of 8 weeks.
  First step: Monotherapy with sertraline (50-200mg). Non responsive patients: 2nd step.
  Second step: Sertraline 200mg + lithium (900mg-1500mg)
  Non responsive patients: 3rd step.
  Third step: Nortriptyline 100mg
  Non responsive patients: 4th step.
  Fourth step: Nortriptyline 100mg + lithium (900mg-1500mg)
  Non responsive patients : 5th step
  Fifth step : Nortriptyline 100mg + sertraline 200mg Non responsive patients
  sixth step: Nortriptyline 100mg + sertraline 200mg + Lithium ( 900mg- 1500mg)
  Interventions: Drug: sertraline; Drug: Nortriptyline; Drug: Lithium

INTERVENTIONS:
Drug: sertraline
  Other Names: Cloridrate of sertraline
Drug: Nortriptyline
  Other Names: Cloridrate of nortrytyline
Drug: Lithium
  Other Names: Lithium Carbonate

SUMMARY:
To evaluate the effectiveness of one algorithm for Major Depression Disorder (MDD) using medications available in the Brazilian Public Healthcare System (SUS), and assessment of the quality of life of these patients.

A randomized pragmatic trial was conducted. An algorithm was developed for the treatment of episodes of unipolar depression episodes.

DETAILED DESCRIPTION:
The study design was that of a pragmatic randomized clinical trial to evaluate the effectiveness of treatments for mood disorders in a public healthcare context in the city of Porto Alegre, in southern Brazil. The algorithm was originally developed for the treatment of major depression by a Delphi panel of experts from psychiatric associations in Brazil. All subjects provided an informed consent form, in writing, in order to participate in the study protocol, which was approved by the institutional ethics committee.

Procedures and measurements of the study

The subjects under evaluation were selected and they followed the stages defined by the treatment protocol:

1. Sample selection by being referred from the primary healthcare clinics in the municipality;
2. Informative talk about mood disorders and the research, with the informed consent forms being provided to the subjects;
3. Screening for unipolar depression episodes with the use of the Patient Health Questionnaire (PHQ-9), and Hypomanic Symptoms Checklist Brazilian Version (HCL -32-BV);
4. Diagnostic evaluation through the Mini International Neuropsychiatric Interview (MINI) and clinical interview for individuals with positive results in the screening instruments;
5. Baseline and demographic assessments using standardized semi-structured interviews in the first and second visits;
6. In each clinic visit, the severity of the symptoms were evealuated using the Clinical Global Impression Scale (CGI), Hamilton Rating Scale for Depression (HRSD), and Young Manic Rating Scale (YMRS);
7. Biweekly follow-up, changed to monthly after stabilization - with a maximum follow-up period of 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. ages between 18 and 65;
2. current acute unipolar depression episode;
3. total capacity to understand and respond to self-applied instruments;
4. the presence of symptoms in the last 30 days;
5. abstinence for at least 30 days for drug addicts

Exclusion Criteria:

1. presence of Organic Brain Syndrome (OBS);
2. pregnancy or lactation;
3. criteria for psychiatric hospitalization.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2010-05; Primary Completion 2014-11 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo Fleck, PhD, Principal Investigator — Federal University of Rio Grande do Sul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lima AF, Miguel SR, Cohen M, Zimmermann JJ, Shansis FM, Cruz LN, Ziegelmann PK, Polanczyk CA, Fleck MP. Effectiveness evaluation of mood disorder treatment algorithms in Brazilian public healthcare patients. Braz J Psychiatry. 2018 Jan-Mar;40(1):26-34. doi: 10.1590/1516-4446-2016-2147. Epub 2017 Aug 21. PMID 28832750

RESULTS

PARTICIPANT FLOW:
Groups:
- Sertraline: Group Started: sertraline (50mg-200mg)
  Subjects evaluated for responsiveness every 2 weeks. Responsive to treatment patients remain in the same step. Max. step duration of 8 weeks.
  First step: Monotherapy with sertraline (50-200mg). Non responsive patients: 2nd step.
  Second step: Sertraline 200mg + lithium (900mg-1500mg)
  Non responsive patients: 3rd step.
  Third step: Nortriptyline 100mg
  Non responsive patients: 4th step.
  Fourth step: Nortriptyline 100mg + lithium (900mg-1500mg)
  Non responsive patients : 5th step
  Fifth step : Nortriptyline 100mg + sertraline 200mg Non responsive patients
  sixth step: Nortriptyline 100mg + sertraline 200mg + Lithium ( 900mg- 1500mg)
  sertraline
  Nortriptyline
  Lithium
Period: Overall Study
Arm/Group | Sertraline
Started | 68
Completed | 43 (Primary and secondary outcomes are assessed just at the end of the protocol, not at each step)
Not Completed | 25

BASELINE CHARACTERISTICS:
Arm/Group | Sertraline
Number analyzed (Participants) | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.4 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53
  Male | 15
Region of Enrollment [Number; unit: participants]
  Brazil | 68

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Response to Treatment
Description: Response to treatment was defined as a 50% reduction from baseline scores in Hamilton Rating Scale for Depression (HRSD). The HRSD is abbreviated version, consists of 17 items. The cutoff points are: 7-17 for mild depression,18-24 for moderate depression, and 25 or more for severe depression .
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Sertraline
Number analyzed (Participants) | 68
Participants | 58

2. Secondary Outcome: Number of Participants With Remission to Treatment
Description: The remission outcome was established as obtaining three consecutive scores of values considered asymptomatic in the Hamilton Rating Scale for Depression (HRSD <7 points) . The subjects that were asymptomatic for at least 6-8 month were considered to be in remission, according to the criteria for partial and complete remission in the DSM-IV.
Time Frame: 8 months
Measure: Count of Participants; unit: Participants
Arm/Group | Sertraline
Number analyzed (Participants) | 68
Participants | 32

3. Secondary Outcome: Quality of Life -WHOQOL Intrument Scores
Description: QOL scores as measured by World Heath Organization Quality of Life - WHOQOL -BREF instrument.
  scores 0-20 . Higher scores means a better outcome. The measure presented is a overall domain with the mean (SD)
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sertraline
Number analyzed (Participants) | 68
score on a scale | 9.45 (3.01)

ADVERSE EVENTS:
Time Frame: 18 months
Arm/Group | Sertraline
Serious Adverse Events (participants affected / at risk) | 0/68
Other Adverse Events (participants affected / at risk) | 0/68

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No